CLINICAL TRIAL: NCT00408070
Title: Phase 2 Study of Bevacizumab in Combination With Carboplatin and Paclitaxel in Patients With Ovarian, Fallopian Tube or Primary Peritoneal Carcinoma
Brief Title: Bevacizumab Study With Carboplatin & Paclitaxel in Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Did not meet accrual goals.
Sponsor: UConn Health (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVF 3696s; IRB 06-337-1
Record Dates: First submitted 2006-12-05; First posted 2006-12-06 (Estimated); Results first posted 2010-11-16 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-02

CONDITIONS: Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer; Stage 3 Cancer; Stage 4 Cancer
Keywords: ovarian cancer; fallopian tube cancer; peritoneal cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Neoplasms | interventions — Bevacizumab; Carboplatin; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I (Experimental): This is a single Arm study. Two of the study drugs used are non-experimental. One of the study drugs is experimental.
  Interventions: Drug: Bevacizumab; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Bevacizumab — cycle 2 (6 cycles re-evaluated and follow up)
  Other Names: Avastin (brand name)
Drug: Carboplatin — cycle #1 and continuous through entire regimen; treated every 3 weeks
  Other Names: Paraplatin
Drug: Paclitaxel — cycle #1 and continuous through entire regimen; treated every 3 weeks
  Other Names: Taxol (brand name)

SUMMARY:
The primary objective is to determine whether the addition of bevacizumab to a regimen of carboplatin plus paclitaxel significantly improves Progression Free Survival (PFS) for patient with Stage III suboptimally cytoreduced or Stage IV ovarian, primary peritoneal or fallopian tube carcinomas.

DETAILED DESCRIPTION:
The aim of this study is to determine if the addition of bevacizumab to a regimen of carboplatin/paclitaxel increases the time to disease recurrence (longer remission for patients) in women that have Stage III suboptimally reduced or Stage IV ovarian cancer.

The hypothesis is that the addition of bevacizumab to a carboplatin/paclitaxel regimen will increase progression free survival in subjects that have Stage III suboptimal cytoreduced or Stage IV ovarian cancer.

Scientific Background and Significance: Vascular endothelial growth factor (VEGF) is found in most tissues, and is known to regulate angiogenesis in both normal (e.g. ovulation) and abnormal (e.g. malignant tumors) conditions. VEGF has been found to be overexpressed in several tumor types, including breast, bladder, uterine, cervical, and relevant to this application, primary and metastatic tumors of patients with advanced ovarian cancer. It is widely believed that the overexpression of this factor contributes to tumorigenesis by supplying a conduit through which oxygen and nutrients can reach and feed the growing malignancy.

Treatment with an anti-VEGF antibody may help to exert a direct anti-angiogenic effect by binding to and clearing VEGF from the tumor microenvironment, thus preventing the formation of new blood vessels. Bevacizumab is a recombinant humanized anti-VEGF monoclonal antibody that inhibits the growth of a number of human cancers, including ovarian cancer. Additional antitumor activity may be obtained through the effects of bevacizumab on tumor vasculature, interstitial pressure, and blood vessel permeability, all of which could allow for enhanced delivery of concurrently administered chemotherapeutic agents to tumor cells.

Based on preliminary data (Proc Am Soc Clin Oncol 2005; 23:A5000 and A 5009), there is biologic rationale to use bevacizumab in the treatment of advanced ovarian cancer. These 2 preliminary studies reported an improved progression-free survival in patients with recurrent ovarian cancer with the use of bevacizumab in combination with chemotherapy. Based on this activity in the recurrent setting, the activity of bevacizumab needs to be evaluated in chemotherapy-naïve patients with advanced ovarian cancer. The purpose of this clinical trial is to determine whether the addition of bevacizumab to a regimen of carboplatin and paclitaxel significantly improves Progression Free Survival (PFS) in patients with Stage III suboptimally cytoreduced or Stage IV ovarian, primary peritoneal or fallopian tube carcinomas.

It is apparent that newer innovative therapies are needed in the front line setting to decrease recurrences and improve survival. The addition of bevacizumab, the anti-vascular endothelial growth factor antibody, to the standard carboplatin/taxol treatment paradigm might help to increase the long-term survival rates in patients newly diagnosed with advanced suboptimal ovarian cancer. The proposed study addresses this issue. The investigational plan that will be utilized to test the hypothesis that the addition of bevacizumab extends the survival time of the affected patients is outlined below.

Women with Stage III or IV ovarian cancer/primary peritoneal cancer/fallopian tube cancer that have undergone surgery with residual suboptimally cytoreduced disease (suboptimal defined as >1cm disease) will be eligible for treatment with one 21-day cycle of carboplatin and paclitaxel and five 21-day cycles of bevacizumab, carboplatin and paclitaxel for a total of six treatment cycles; bevacizumab treatment is delayed by one cycle to ensure adequate post-surgical healing. Subjects will be evaluated by CT scans to determine response to therapy; individuals that progress will be withdrawn from the study. The CT scan conducted after the completion of therapy will dictate the next course of action. Patients demonstrating a complete response will be maintained on bevacizumab as consolidation therapy; subjects demonstrating a partial response will continue to receive bevacizumab, carboplatin and paclitaxel. The total treatment time for patients with a clinical response following the initial 6 cycles of therapy will be 12 months. Prior to starting consolidation therapy, all patients with a complete clinical response or in those for whom surgery may result in a complete secondary cytoreduction, will be given the option of undergoing a second look surgery. The findings at surgery in combination with the CT scan will determine the response to initial therapy. The decision not to participate in the second look surgery will not affect the follow-up treatment that the patient will receive.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of primary peritoneal carcinoma, fallopian tube epithelial ovarian carcinoma,
* stage III suboptimal surgery or biopsy,
* stage IV disease
* no prior chemotherapy

Exclusion Criteria:

* unstable heart conditions
* high blood pressure
* vascular disorders
* bleeding problems

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-10; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Runowicz, MD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab Plus Carboplatin and Paclitaxel: This is a single Arm study. Two of the study drugs used are non-experimental. One of the study drugs is experimental.Cycle one - Paclitaxel 175 mg/m2 iv; Carboplatin AUC 6 iv; Cycle two through six - Paclitaxel 175 mg/m2 iv; Carboplatin AUC 6 iv; Avastin 15 mg/kg IV Repeat cycle every 21 days, total of 6 cycles
Period: Overall Study
Arm/Group | Bevacizumab Plus Carboplatin and Paclitaxel
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab Plus Carboplatin and Paclitaxel
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (11.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival Rate at 9 Months
Description: This Outcome is measuring the number of particpants who have survived.
Time Frame: 9 months
Measure: Number; unit: participants
Arm/Group | Bevacizumab Plus Carboplatin and Paclitaxel
Number analyzed (Participants) | 5
participants | 4

2. Secondary Outcome: Response to Treatment (Clinical/Pathological)
Time Frame: 12 months
Population: not assessed; study terminated early
Arm/Group | Bevacizumab Plus Carboplatin and Paclitaxel
Number analyzed (Participants) | 0

3. Secondary Outcome: Rate of Decline of CA-125
Time Frame: 12 months
Population: not assessed; study terminated early
Arm/Group | Bevacizumab Plus Carboplatin and Paclitaxel
Number analyzed (Participants) | 0

4. Secondary Outcome: To Determine the Degree and Type of Toxicity of This Combined Regimen
Time Frame: weekly
Population: not assessed; study terminated early
Arm/Group | Bevacizumab Plus Carboplatin and Paclitaxel
Number analyzed (Participants) | 0

5. Secondary Outcome: Determine Tolerability to 12 Months (q 3 Weeks) of Bevacizumab Maintenance Therapy
Time Frame: 12 months
Population: not assessed; study terminated early
Arm/Group | Bevacizumab Plus Carboplatin and Paclitaxel
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Bevacizumab Plus Carboplatin and Paclitaxel
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab Plus Carboplatin and Paclitaxel (N=5)
Neuropathy - motor (Nervous system disorders) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab Plus Carboplatin and Paclitaxel (N=5)
hemoglobin decrease (Blood and lymphatic system disorders) | 5
alopecia (Skin and subcutaneous tissue disorders) | 2
pain - musculoskeletal; joint (Musculoskeletal and connective tissue disorders) | 2
arthritis (Musculoskeletal and connective tissue disorders) | 1
allergic reaction / hypersensitivity (Immune system disorders) | 2
bloating /abdominal distention (Gastrointestinal disorders) | 1
metabolic laboratory - other (Blood and lymphatic system disorders) | 1 — elveated BUN/Creatinine
bruising (Skin and subcutaneous tissue disorders) | 1
confusion (Nervous system disorders) | 1
constipation (Gastrointestinal disorders) | 2
dehydration (Gastrointestinal disorders) | 2
diarrhea (Gastrointestinal disorders) | 3
dysgeusia (Gastrointestinal disorders) | 3
metabolic laboratory - other (Blood and lymphatic system disorders) | 1 — AST,ALT decreased
dizziness (Nervous system disorders) | 1
edema - limb (Blood and lymphatic system disorders) | 1
alkaline phosphatase - elevated (Blood and lymphatic system disorders) | 1
creatinine - elevated (Blood and lymphatic system disorders) | 2
ALT (SGPT) - evelated (Blood and lymphatic system disorders) | 1
AST (SGOT) - elevated (Blood and lymphatic system disorders) | 1
lactose dehydrogenase (LDH) - elevated (Blood and lymphatic system disorders) | 1
fatigue (General disorders) | 5
febrile neutorpenia (Infections and infestations) | 1
flatulence (Gastrointestinal disorders) | 1
gastritis (Gastrointestinal disorders) | 1
dyspepsia (Gastrointestinal disorders) | 3
headache (General disorders) | 1
hearing alteration (Ear and labyrinth disorders) | 1
hemoglobin - elevated (Blood and lymphatic system disorders) | 1
hyperglycemia (Metabolism and nutrition disorders) | 4
hypoalbuminemia (Blood and lymphatic system disorders) | 4
hyponatremia (Blood and lymphatic system disorders) | 5
hypocalcemia (Blood and lymphatic system disorders) | 2
hypokalemia (Blood and lymphatic system disorders) | 1
hypomagnesemia (Blood and lymphatic system disorders) | 4
hypertension (Cardiac disorders) | 2
Infection - skin (Infections and infestations) | 1
infection - urinary tract (Infections and infestations) | 2
infection - upper respiratory (Infections and infestations) | 2
infection - NOS (Infections and infestations) | 1
injection site reaction (Skin and subcutaneous tissue disorders) | 1
leukocytes - decreased (Blood and lymphatic system disorders) | 5
bicarbonate - decreased (Blood and lymphatic system disorders) | 2
pain, bone (Musculoskeletal and connective tissue disorders) | 1
lymphopenia (Blood and lymphatic system disorders) | 3
mucositis/stomatitis (Gastrointestinal disorders) | 1
memory impairment (Nervous system disorders) | 1
muscle weakness (Musculoskeletal and connective tissue disorders) | 1
nasal/sinus reactions (Respiratory, thoracic and mediastinal disorders) | 3
nail changes (Skin and subcutaneous tissue disorders) | 1
nausea (Gastrointestinal disorders) | 4
neuropathy - sensory (Nervous system disorders) | 5
neuropathy - cranial (Nervous system disorders) | 1
neutrophils/granulocytes - decreased (Blood and lymphatic system disorders) | 5
pain - extremity (Musculoskeletal and connective tissue disorders) | 2
pain - muscle (Musculoskeletal and connective tissue disorders) | 1
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
proteinuria (Renal and urinary disorders) | 2
pruritus (Skin and subcutaneous tissue disorders) | 1
rigors / chills (General disorders) | 1
rash (Skin and subcutaneous tissue disorders) | 1
eczema (Skin and subcutaneous tissue disorders) | 1
allergic rhinitis (Immune system disorders) | 1
platelets - decreased (Blood and lymphatic system disorders) | 5
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
vomiting (Gastrointestinal disorders) | 3
dysarthria (Respiratory, thoracic and mediastinal disorders) | 1
weight loss (Metabolism and nutrition disorders) | 1
neuropathy - cranial -CN V (Nervous system disorders) | 1
respiratory - other (cold symptoms) (Respiratory, thoracic and mediastinal disorders) | 1
seroma (Musculoskeletal and connective tissue disorders) | 1

LIMITATIONS AND CAVEATS:
This trial ended early after enrolling only 5 of 100 patients. Due to the small enrollment number and incomplete data set, no data analyses were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less